CLINICAL TRIAL: NCT06660823
Title: Role of Levothyroxine Supplementation in Delayed Recovery Following Cardiac Surgery
Acronym: L-Thyroxine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, sarah hamdy, Lecturer of Anesthesia,ICU and pain management, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU R237/2024
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Results first posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Cardiac Surgery Intensive Care Treatment; Delayed Recovery From Anaesthesia; Euthyroid Sick Syndrome; Cardiac Surgery Requiring Cardiopulmonary Bypass
Keywords: L-Thyroxine; Delayed recovery post cardiac surgery; hypthyroidism
MeSH Terms: conditions — Delayed Emergence from Anesthesia; Euthyroid Sick Syndromes | interventions — Thyroxine

STUDY DESIGN:
Intervention Model Description: This study is a prospective, randomized controlled trial that will study the postoperative clinical outcomes of levothyroxine supplementation in delayed recovery or prolonged ventilation patients post cardiac surgery.
  Randomization will be performed using a computer-generated randomization sequence and allocation concealment to be maintained all through the time of procedure, by using opaque, numbered, and sealed envelopes.
  Patients will be randomly allocated by computer generated randomization into two groups A and B:
  * Group A (Study group): patients receiving oral supplementation of levothyroxine.
  * Group B (Control): patients receiving Placebo drug.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Study group) (Active Comparator): group A will receive levothyroxine via Ryle, dose of 25 to 50 ug/ day according to BMI
  Interventions: Drug: L-thyroxine
- Group B (Control) (Placebo Comparator): group B will receive placebo in form of inert starch tablet
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: L-thyroxine — Patients who show signs of delayed recovery defined as either prolonged ventilation for 48 hours or delayed conscious level recovery for 48 hours despite exclusion of muscle relaxants and/or sedative drugs. Those patients will undergo CT brain, CT chest and neurological examination to exclude structural damage as per institutional protocols. Also, metabolic profile screening including full kidney function, full liver function, electrolyte to exclude correctable metabolic abnormalities. and thyroid profile (TSH, free T3, free T4) sick euthyroid patients who are having normal FreeT3, normal Free T4, low TSH and low level of free T3 or freeT4 will be included in the study according lab reference.Daily assessment of conscious level according to Glasgow Coma Scale (GCS) and spontaneous breathing trial by ICU consultant (the investigator) till ICU discharge.
  Patients will receive levothyroxine via Ryle, dose of 25 to 50 ug/ day according to BMI.
  Arms: Group A (Study group)
Drug: Placebo Oral Tablet — patients will receive placebo oral tablet
  Arms: Group B (Control)

SUMMARY:
Research indicates that hypothyroidism decreases heart contractility, reduces stroke volume and rate, affects the vascular endothelium, and increases the risk of atherosclerosis, systemic vascular resistance, hypertension, atherogenic lipid profile, and coagulation abnormality .

Hypothyroidism was reported to be strongly related to cardiovascular disease, respiratory complications, neurological complications, and a significant difference in ventilator weaning time.

Once subclinical hypothyroidism patients are treated with levothyroxine, their physical fitness measured by a 6-minute walk is significantly improved, also showed that levothyroxine treatment can optimize the treatment of heart failure with preserved functions (HFpEF) and heart failure with reduced functions (HFrEF) patients with systolic left ventricular dysfunction and sub clinical hypothyroidism (SCH).

The primary aim of this study is to investigate the effect of supplementation of oral levothyroxine in delayed recovery patients post cardiac surgery.

DETAILED DESCRIPTION:
Research indicates that hypothyroidism decreases heart contractility, reduces stroke volume and rate, affects the vascular endothelium, and increases the risk of atherosclerosis, systemic vascular resistance, hypertension , atherogenic lipid profile, and coagulation abnormality .

Hypothyroidism was reported to be strongly related to cardiovascular disease, respiratory complications, neurological complications, and a significant difference in ventilator weaning time. Severe thyroid dysfunction is related to muscle relaxation and lead to respiratory muscle depression and disturbed conscious level.Surgical stress of cardiac surgery might be followed by a prolonged recovery process and cardiac dysfunction .

The exact physiology of thyroid disease and the relationship with post cardiac surgery remain unclear. Thus far, large-scale clinical statistical analysis evidence on the complication rate and long-term mortality is lacking. Current important prognostic assessment tools such as EuroSCORE II , and Society of Thoracic Surgeons (STS) score do not include thyroid function assessment, even though it has a significant impact on the metabolic, cardiovascular, and circulation system.

Once subclinical hypothyroidism patients are treated with levothyroxine, their physical fitness measured by a 6-minute walk is significantly improved, also showed that levothyroxine treatment can optimize the treatment of heart failure with preserved functions (HFpEF) and heart failure with reduced functions (HFrEF) patients with systolic left ventricular dysfunction and sub clinical hypothyroidism (SCH).

The heart is a major target of thyroid hormones, with maintenance of euthyroid hormone balance critical for proper function. Moreover, thyroid hormones have been shown a vital role in cardiac repair after injury beyond their roles in development and metabolism homeostasis.

After cardiac surgery with cardiopulmonary bypass (CPB), however, serum thyroid hormone levels are often decreased, especially in pediatric patients. This is called as the euthyroid sick syndrome (ESS).

It is reported that after cardiac surgery with CPB, 50% to 75% of adult patients present a decreased serum level of triiodothyronine (T3) (type 1 ESS) and 100% of pediatric patients display decreased serum levels of both T3 and tetraiodothyronine (T4) (type 2 ESS).

Because ESS has been associated with increased morbidity after cardiac surgery, it is deemed that intravenous supplementation of thyroid hormones in postoperative period is benefit to infants and small children. This view is supported by the largest randomized clinical trial so far, the Triiodothyronine for Infants and Children Undergoing CPB (TRICC) study, in which subgroup analysis shows a significant reduction in mechanical ventilation time, less use of inotropic drugs, and better cardiac function with intravenous T3 supplementation after surgery in pediatric patients aged <5 months.

Ischemia and reperfusion occur during almost every cardiac surgery and myocardial ischemia/reperfusion injury (IRI) is an important cause of morbidity and mortality in the early postoperative period after cardiac surgery. It has been shown that thyroid hormones can limit myocardial IRI via a fine balance between proapoptotic and prosurvival signaling pathways.Furthermore, thyroid hormones can provide a protection against myocardial IRI by inducing pharmacological preconditioning.The available evidence also indicates that perioperative oral T3 therapy can significantly attenuate the postoperative decline in serum T3 level or maintain total and free serum T3 levels within normal limits in adult and pediatric patients undergoing cardiac surgery.Given that oral administration is a safe, convenient and feasible route of perioperative medication. This has been proven by the single-center, prospective, double blind, randomized placebo-controlled clinical pilot trial including 40 patients receiving a dose of 0.4mg/kg (trial group, thyroid tablet taken orally once a day, for 4 days before surgery).In summary, this pilot study demonstrated that children after cardiac surgery with CPB are at a high risk to develop postoperative ESS. Preoperatively short-term oral thyroid hormones can reduce severity of postoperative ESS without negative effects and provides a protection against myocardial IRI by increasing HSP70 and MHCa expression.

In another reported double blind, placebo-controlled trial in 100 infants with normal thyroid function. Subjects underwent cardiac surgery and were randomly assigned during a 16-month period into 2 groups (50 in the thyroxine supplementation group and 50 in the placebo group) to determine whether there was an association between oral thyroxine (T4) supplementation and changes in cardiac index (CI), along with other important outcomes. Subjects in the study group received an oral dose of 5 µg/kg of T4 starting 12 hours before surgery and every morning thereafter while in the intensive care unit. Subjects in the study group had higher CI than did the placebo group (CI 0.30 L/min/m2 higher; P = .04).

It has been well described that early after the initiation of CPB, particularly DHCA, thyroid-stimulating hormone concentration is raised, responding to decreased concentrations of triiodothyronine (T3), and that levels restore during a period of days, beginning with thyroid stimulating hormone and followed by T3, an entity referred as ''euthyroid sick syndrome.'' An actual etiology for these changes has not been precisely described; however, hemodilution, hypothermia, and inflammation have been implicated. As of now, thyroid hormone supplementation remains the mainstay therapy for euthyroid sick syndrome.

This study , like several others, demonstrates that perioperative thyroid hormone supplementation is associated with improved outcomes. They demonstrated that Thyroid hormone levels are reduced significantly in the immediate postoperative period after open-heart surgery. Oral T4 supplementation improves the CI and reduces the inotropic requirement. In addition, it reduces the duration of mechanical ventilation, ICU and hospital stay, and TISS in infants after surgery for complex congenital heart defects.

Routinely, patients with delayed recovery and/or prolonged mechanical ventilation are managed as follow :

1. Full neurological examination, CT brain, repeated CT brain after 48-hour, MRI stroke protocol, adding of brain stimulants medications and if fits developed antiepileptics would be added accordingly.
2. Liver profile checked and liver support added,
3. Renal profile checked, stoppage of nephrotoxic drugs, fluids chart, renal dose adjustment of medications.
4. Blood sugar hourly monitored.
5. Sepsis surveillance by withdrawing pan cultures, replacing old IV catheters upgrading antibiotics accordingly.

This is typically included in institutional ICU protocol. The primary aim of this study is to investigate the effect of supplementation of oral levothyroxine in delayed recovery patients post cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* • Age group: Adult patients from age of 45 to70 years. (Majority of our patients falls in this age group 45-70 years, below these patients are relatively young and usually do not show delayed recovery or prolonged ventilation, while above 70 years are considered frail and more vulnerable to anesthetic medications, so we preferred to exclude them)

  * Sex: Both sexes
  * Elective, urgent and emergency open heart surgeries. (Most of urgent and emergency cases are either mechanical valve thrombosis or aortic dissection patients, and are more prone to prolonged mechanical ventilation and delayed recovery compared to elective patients)

Exclusion Criteria:

* • Patients refuse to give informed consent.

  * Patient younger than 45 years old, older than 70 years old.
  * Off pump patients.
  * Patients known hypothyroidism on levothyroxine supplementation.
  * Patients known hyperthyroidism on Carbimazole.
  * Those developing any form of arrhythmia L-Thyroxine will be stopped immediately and the patient will be excluded from the study.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-11-30 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine ,Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Duntas LH, Jonklaas J. Levothyroxine Dose Adjustment to Optimise Therapy Throughout a Patient's Lifetime. Adv Ther. 2019 Sep;36(Suppl 2):30-46. doi: 10.1007/s12325-019-01078-2. Epub 2019 Sep 4. PMID 31485977
- [Background] Flores S, Checchia PA. Inflammatory and neurohormonal modulation for congenital heart surgery: The quest continues. J Thorac Cardiovasc Surg. 2018 Sep;156(3):1207-1208. doi: 10.1016/j.jtcvs.2018.06.004. Epub 2018 Jun 22. No abstract available. PMID 30005886
- [Background] Batra YK, Singh B, Chavan S, Chari P, Dhaliwal RS, Ramprabu K. Effects of cardiopulmonary bypass on thyroid function. Ann Card Anaesth. 2000 Jul;3(2):3-6. PMID 17848764
- [Background] Zhang JQ, Yang QY, Xue FS, Zhang W, Yang GZ, Liao X, Meng FM. Preoperative oral thyroid hormones to prevent euthyroid sick syndrome and attenuate myocardial ischemia-reperfusion injury after cardiac surgery with cardiopulmonary bypass in children: A randomized, double-blind, placebo-controlled trial. Medicine (Baltimore). 2018 Sep;97(36):e12100. doi: 10.1097/MD.0000000000012100. PMID 30200092
- [Background] Kumar A, Taliyan R, Sharma PL. Evaluation of thyroid hormone induced pharmacological preconditioning on cardiomyocyte protection against ischemic-reperfusion injury. Indian J Pharmacol. 2012 Jan;44(1):68-72. doi: 10.4103/0253-7613.91870. PMID 22345873
- [Background] Plumpton K, Haas NA. Identifying infants at risk of marked thyroid suppression post-cardiopulmonary bypass. Intensive Care Med. 2005 Apr;31(4):581-7. doi: 10.1007/s00134-004-2549-1. Epub 2005 Jan 28. PMID 15678312
- [Background] Gerdes AM, Ojamaa K. Thyroid Hormone and Cardioprotection. Compr Physiol. 2016 Jun 13;6(3):1199-219. doi: 10.1002/cphy.c150012. PMID 27347890
- [Background] Biondi B, Klein I. Hypothyroidism as a risk factor for cardiovascular disease. Endocrine. 2004 Jun;24(1):1-13. doi: 10.1385/ENDO:24:1:001. PMID 15249698

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A (Study Group): group A will receive levothyroxine via Ryle, dose of 25 to 50 ug/ day according to BMI
  L-thyroxine: Patients who show signs of delayed recovery defined as either prolonged ventilation for 48 hours or delayed conscious level recovery for 48 hours despite exclusion of muscle relaxants and/or sedative drugs. Those patients will undergo CT brain, CT chest and neurological examination to exclude structural damage as per institutional protocols. Also, metabolic profile screening including full kidney function, full liver function, electrolyte to exclude correctable metabolic abnormalities. and thyroid profile (TSH, free T3, free T4) sick euthyroid patients who are having normal FreeT3, normal Free T4, low TSH and low level of free T3 or freeT4 will be included in the study according lab reference.Daily assessment of conscious level according to Glasgow Coma Scale (GCS) and spontaneous breathing trial by ICU consultant (the investigator) till ICU discharge.
  Patients will receive levothyroxine via Ryle, dose of 25 to 50 ug/ day according to BMI.
Period: Overall Study
Arm/Group | Group A (Study Group) | Group B (Control)
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A (Study Group) | Group B (Control) | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.94 (15.33) | 57.57 (7.12) | 55.76 (12.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 11 | 28
  Male | 18 | 24 | 42
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Glasgow Coma Scale (GCS) From Intervention Initiation to ICU Discharge (Δ)
Description: The Glasgow Coma Scale (GCS) assesses conscious level through three components:
  Eye response (scored 1-4):
  4: Opens eyes spontaneously
  3: Opens eyes to verbal command
  2: Opens eyes to pain
  1: No eye opening
  Verbal response (scored 1-5):
  5: Oriented and converses
  4: Confused
  3: Inappropriate words
  2: Incomprehensible sounds
  1: No verbal response
  Motor response (scored 1-6):
  6: Obeys commands
  5: Localizes to pain
  4: Withdraws from pain
  3: Abnormal flexion (decorticate)
  2: Abnormal extension (decerebrate)
  1: No motor response
  The total GCS score ranges from 3 (worst) to 15 (best), with higher scores indicating better neurological function. The primary outcome is the change in total GCS score from baseline (48 hours postoperatively, before intervention) to ICU discharge.
Time Frame: From intervention initiation (48 hours postoperatively) to ICU discharge, up to 1 month postoperatively. (i.e., within 28 days after baseline).
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Group A (Study Group) | Group B (Control)
Number analyzed (Participants) | 35 | 35
Score on a scale | 6.65 (3.60) | 2.69 (0.64)

2. Secondary Outcome: Total Duration of Mechanical Ventilation
Description: Total time (in hours) from initiation of mechanical ventilation postoperatively until successful extubation, including time before and after study intervention.
Time Frame: From surgery completion until extubation (assessed for ≤30 days postoperatively).
Population: All 70 participants included in intention-to-treat analysis. Duration calculated for survivors until extubation; deceased patients contributed ventilation hours until death.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Group A (Study Group) | Group B (Control)
Number analyzed (Participants) | 35 | 35
hours | 130.40 (75.74) | 142.14 (41.37)

3. Secondary Outcome: Duration of Intensive Care Unit (ICU) Stay
Description: Total time (in days) from ICU admission after cardiac surgery until discharge from ICU or death.
Time Frame: From ICU admission until discharge/death (assessed for ≤30 days postoperatively).
Population: All 70 participants included in intention-to-treat analysis. Duration calculated for:
  Survivors: Until ICU discharge
  Non-survivors: Until death in ICU
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group A (Study Group) | Group B (Control)
Number analyzed (Participants) | 35 | 35
days | 9.03 (5.42) | 7.51 (1.80)

4. Secondary Outcome: Total Hospital Stay Stay.
Description: The total hospital stay will be recorded in days and compared between both groups.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group A (Study Group) | Group B (Control)
Number analyzed (Participants) | 35 | 35
days | 13.06 (4.49) | 10.29 (3.48)

5. Secondary Outcome: Average Inotropic Support Infusion Rate in ICU
Description: Average infusion rate (in ng/kg/min) of norepinephrine and epinephrine administered during ICU stay. Calculated as total dose (ng) divided by patient weight (kg) and total infusion duration (minutes). Does not include intraoperative inotropic support.
Time Frame: From ICU admission until discontinuation of inotropic support or ICU discharge (assessed daily for ≤30 days).
Population: All 70 participants were included in the analysis per intention-to-treat. Average infusion rates were calculated based on the total dose administered, patient weight, and total duration of infusion during the ICU stay.
Measure: Mean (Standard Deviation); unit: ng/kg/min
Arm/Group | Group A (Study Group) | Group B (Control)
Number analyzed (Participants) | 35 | 35
ng/kg/min
  Nor Epinephrine | 79.60 (51.60) | 135.86 (93.98)
  Epinephrine | 83.70 (40.21) | 137.93 (78.26)

6. Secondary Outcome: Change in Left Ventricular Ejection Fraction (LVEF) From Baseline to ICU Discharge
Description: Absolute change in left ventricular ejection fraction (LVEF) measured by transthoracic echocardiography, calculated as:
  Δ EF = Postoperative EF
  - Preoperative EF Δ EF
  * Postoperative EF-Preoperative EF Negative values indicate decline in cardiac function.
Time Frame: Preoperative assessment: Within 24 hours before surgery Postoperative assessment: At ICU discharge (≤30 days postoperatively)
Population: All 70 participants included in intention-to-treat analysis. Echocardiography performed by blinded cardiologists per institutional protocols.
Measure: Mean (Standard Deviation); unit: Percentage points of ejection fraction
Arm/Group | Group A (Study Group) | Group B (Control)
Number analyzed (Participants) | 35 | 35
Percentage points of ejection fraction | -6.15 (4.32) | -19.14 (10.21)

7. Secondary Outcome: Number of Participants With New-onset Supraventricular Arrhythmia
Description: Incidence of new-onset supraventricular arrhythmias (atrial fibrillation, atrial flutter, or supraventricular tachycardia) confirmed by 12-lead ECG during ICU stay. Excludes pre-existing arrhythmias.
Time Frame: From ICU admission until discharge or death (≤30 days postoperatively).
Population: All 70 participants included in intention-to-treat analysis. Arrhythmias diagnosed by blinded cardiologists using:
  Continuous ECG monitoring
  12-lead ECG for confirmation
Measure: Number; unit: participants
Arm/Group | Group A (Study Group) | Group B (Control)
Number analyzed (Participants) | 35 | 35
participants | 1 | 13

ADVERSE EVENTS:
Time Frame: 30 day
Description: adverse events were already defined as all cause mortality and arrhythmias
Arm/Group | Group A (Study Group) | Group B (Control)
All-Cause Mortality (participants affected / at risk) | 5/35 | 16/35
Serious Adverse Events (participants affected / at risk) | 1/35 | 13/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (Study Group) (N=35) | Group B (Control) (N=35)
Arrhythmias (Cardiac disorders) | 1 (1) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-01): https://cdn.clinicaltrials.gov/large-docs/23/NCT06660823/Prot_SAP_000.pdf